CLINICAL TRIAL: NCT05688124
Title: A Randomized, Open-label, Two-cycle Clinical Study to Evaluate the Drug Interaction, Food Effect and Pharmacokinetics of IBI351 With Esomeprazole in Healthy Subjects
Brief Title: A Study of IBI351 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIBI351P001
Record Dates: First submitted 2022-12-12; First posted 2023-01-18 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI351 (Other): This cohort investigated the effect of food on the pharmacokinetics of IBI351 in healthy subjects. In a double-crossover design, subjects were enrolled and randomly divided into two test groups A and B. Group A: IBI351 was orally administered to subjects in this group on an empty stomach on Day 1, followed by a high-fat meal on Day 4. Group B: IBI351 was orally administered to subjects in this group after a high-fat meal on Day 1 followed by an empty stomach on Day 4.
  Interventions: Drug: IBI351
- IBI351+Esomeprazole (Other): Enrolled subjects were orally administered IBI351 with recommended dose on an empty stomach. Esomeprazole were administered orally.
  Interventions: Drug: IBI351; Drug: Esomeprazole

INTERVENTIONS:
Drug: IBI351 — IBI351 is administered orally
Drug: Esomeprazole — Esomeprazole is administered orally
  Arms: IBI351+Esomeprazole

SUMMARY:
This is a randomized, open-label, two-cycle clinical study to evaluate the drug interaction, food effect and pharmacokinetics of IBI351 and esomeprazole in healthy subjects. A total of two cohorts were planned to be enrolled in each cohort. Cohort 1: This cohort investigated the effect of esomeprazole on the pharmacokinetics of IBI351 in healthy subjects. Cohort 2: This cohort investigated the effect of food on the pharmacokinetics of IBI351 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily sign the informed consent form before the trial, fully understand the content, process and possible adverse reactions of the trial, and be able to complete the study according to the requirements of the trial protocol.
2. healthy male subjects aged 18 to 45 years (including both ends) at the time of signing informed consent.
3. body weight is not less than 50 kg, and body mass index (BMI) is within the range of 19 ~ 26 kg/m2 (including cut-off value).

Exclusion Criteria:

1. have taken any products containing alcohol or have a positive alcohol breath test (≥ 20 mg/100 ml) within 24 hours before taking study medication.
2. hepatitis B surface antigen HBsAg positive.
3. hepatitis C virus antibody positive.
4. positive AIDS antigen/antibody or Treponema pallidum antibody

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
maximum concentrations (Cmax ) for plasma | approximately 10 days after first dose
area under the curve from time 0 to infinity(AUC0-inf) for plasma | approximately 10 days after first dose
area under the curve from time 0 to the last time point (AUC0-t) for plasma | approximately 10 days after first dose

SECONDARY OUTCOMES:
time-to-maximum concentration (Tmax) for total plasma | approximately 10 days after first dose
half-life (t1/2) for total plasma | approximately 10 days after first dose
apparent clearance (CL/F) for total plasma | approximately 10 days after first dose
the time prior to the first measurable (non-zero) concentration （tlag） | approximately 10 days after first dose
apparent volume of distribution(Vz/F) for total plasma | approximately 10 days after first dose
adverse events | approximately 10 days after first dose
number of participants with abnormal ECG readings | approximately 10 days after first dose
number of participants with abnormal hematology test results | approximately 10 days after first dose
number of participants with abnormal chemisty test results | approximately 10 days after first dose
number of participants with abnormal vital signs | approximately 10 days after first dose
number of participants with abnormal physical examination | approximately 10 days after first dose

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China